CLINICAL TRIAL: NCT02411669
Title: Effectiveness and Determinants of Effectiveness of Implementation of Tools for the Development of Patient Centred Care at Hospital
Brief Title: Impact of Tools for the Development of Patient Centered Care at Hospital
Acronym: MoSTRA
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2013/32
Record Dates: First submitted 2015-03-27; First posted 2015-04-08 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Patient Centred Care
Keywords: Patient centred care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Health care professionals: Physicians, nurses and managerial staff
  Interventions: Other: Operational patient centered care tools

INTERVENTIONS:
Other: Operational patient centered care tools — The FORAP (Fédération des Organismes Régionaux et territoriaux pour l'Amélioration des Pratiques et des organisations) and the la HAS (High Authority of Health) have developed and validated five tools promoting patient centered care at hospital.
  They can be implemented one by one or in association according to hospital situation. Hospitals should identify the association of tools fitting the most to their objectives and the actions already done.

SUMMARY:
A national context for patient centered care development exists in France at hospital with strong support for the implementation of operational patient centered care tools. Patient centered care is a global vision of patient or family management promoting the respect of patient freedom, of patient listening and of patient needs. Patient centered care is an important issue of quality and security of care. The FORAP (Fédération des Organismes Régionaux et territoriaux pour l'Amélioration des Pratiques et des organisations) and the la HAS (High Authority of Health) have developed and validated five tools promoting patient centered care at hospital.

They can be implemented one by one or in association according to hospital situation. Hospitals should identify the association of tools fitting the most to their objectives and the actions already done.

The objectives of the project are to analyse the effectiveness of the implementation of HAS - FORAP tools on the development of patient centred care at hospital and to analyse the individual and organisational determinants of their effectiveness. It focuses on acute care hospitals that have the choice of the combination of tools and that are followed during two years with combined quantitative and qualitative analyses. Quantitative assessment are based on validated indicators on patient satisfaction, patient centred care development and organizational context. Qualitative data collection are realised in each included hospital and combine individual interviews and focus groups including Physicians, nurses and managerial staff.

ELIGIBILITY:
No specific eligibility criteria for health care professionals

Eligibility criteria for patients:

Inclusion Criteria:

* Patients hospitalized for a minimum of 2 consecutive nights
* Patients contact details known after hospitalization end

Exclusion Criteria:

* Anonymous patient
* Patient deceased during hospitalization
* Patient non resident in France

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are 2 populations participating in this trials:
  * Health care professionals : physicians, nurses and managerial staff
  * Patients
Sampling Method: Non-Probability Sample
Enrollment: 950 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Self assessment score of patient centred care at hospital by health care professionals and patients | At study start in hospital, between 2 to 4 months before tool implementation
Self assessment score of patient centred care at hospital by health care professionals and patients | 6 months after tool implementation for promoting patient centered care at hospital
Self assessment score of patient centred care at hospital by health care professionals and patients | 18 months after tool implementation for promoting patient centered care at hospital

SECONDARY OUTCOMES:
Patients global satisfaction score | At study start, between 2 to 4 months before tool implementation for promoting patient centered care at hospital, 6 month and 18 month after

CONTACTS AND LOCATIONS:
Locations (30):
- France (30):
  - CH d'Agen, Agen
  - Clinique du Parc, Autun
  - CHU de Bordeaux, Bordeaux
  - Maison de santé Marie Galène, Bordeaux
  - Centre François Baclesse, Caen
  - CHU de Caen, Caen
  - Hôpital Privé Saint Martin, Caen
  - CH de Chambéry, Chambéry
  - CH de Crest, Crest
  - Clinique Saint Vincent, Dax
  - CH de Dinan, Dinan
  - Centre orthopédique médico-chirurgical, Dracy
  - CH de Givors, Givors
  - CH de Guingamp, Guingamp
  - CH de Joigny, Joigny
  - CHD de La Roche Sur Yon, La Roche-sur-Yon
  - Clinique Saint Charles, La Roche-sur-Yon
  - Clinique Saint Anne, Langon
  - CH Côte de Lumière, Les Sables-d'Olonne
  - Clinique du Parc, Lyon
  - Clinique du Val d'Ouest, Lyon
  - CH du Haut-Bugey, Oyonnax
  - CH intercommunal de Quimper, Quimper
  - CH de Redon, Redon
  - CHU de Rennes, Rennes
  - CH de St Brieuc, Saint-Brieuc
  - Polyclinique Côte Basque Sud, Saint-Jean-de-Luz
  - Clinique du Parc, Saint-Priest-en-Jarez
  - CH de Vannes, Vannes
  - CH de Vitré, Vitré